CLINICAL TRIAL: NCT03603210
Title: Outcomes of Drug Coated Balloon Angioplasty, A UK Real Life Experience From 2009 to 2015
Acronym: DCBNORWICH
Status: Active, not recruiting | Type: Observational
Sponsor: Julie Dawson (Other)
Responsible Party: Sponsor-Investigator, Julie Dawson, Research Services Manager, Norfolk and Norwich University Hospitals NHS Foundation Trust
Organization: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Other Study IDs: 195002 (167-10-15); NCT04482972 (obsolete NCT alias)
Record Dates: First submitted 2017-11-01; First posted 2018-07-27 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Ischaemic Heart Disease
Keywords: Ischaemic heart disease; coronary angioplasty; drug coated balloons (DCB)
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated with DCB angioplasty: Patient cohort is comprised of all patients who received drug coated balloon angioplasty at NNUH during the above period. Within this cohort there will be two main groups which are drug coated balloon (DCB) angioplasty for de novo coronary artery disease (CAD) and DCB angioplasty for ISR/ST. Graft cases will be reported as a small third group.
  Outcomes will also be reported for three sub groups of de novo disease group, namely, dcb-only angioplasty for de novo disease, dcb-only angioplasty as primary percutaneous coronary intervention (PPCI) and dcb-only angioplasty group using a DCB with a diameter of 3mm or more in de novo disease.
  Interventions: Device: Drug coated balloon angioplasty

INTERVENTIONS:
Device: Drug coated balloon angioplasty — Drug coated balloons are semi compliant percutaneous coronary angioplasty balloons coated with a chemotherapeutic drug such as Paclitaxel used with an excipient which allows rapid absorption to vessel wall upon balloon expansion for 30-60s. This allows coronary angioplasty without any permanent or semi- permanent stent or scaffold provided there are no vessel threatening dissections or significant acute recoil.
  Other Names: DCB

SUMMARY:
This is a single center, retrospective, observational cohort study to assess the safety and efficacy of drug coated balloon (DCB) angioplasty in all forms of coronary artery disease. The Investigators intend to report outcomes of all patients who received DCB angioplasty at their center during the above mentioned period for up to 10 years.

DETAILED DESCRIPTION:
The Investigators expect to assess outcomes of all patients who received Drug Coated Balloon Angioplasty treatment, which is a novel therapy as opposed to standard Drug Eluting Stent insertion, for all types of coronary artery disease from 01/01/2009 till 31/12/2015 in their center. The Investigators believe the number exceeds 1000 patients.

The Investigators plan to collect demographic and procedural data from their existing data base. They will request up to date follow-up events from NICOR (National Institute for Cardiovascular Outcomes Research, UK) in 2017(data ending December 2016), by which time all patientswould have had minimum of 12 months follow up. The Investigators plan to incorporate these findings to their data set and report the comprehensive outcomes. Primary end point will be major adverse cardiac outcomes (MACE) defined as a composite of death, myocardial infarction and target vessel revascularisation. Secondary end points will be acute vessel closure and target lesion revascularisation. The Investigators also have a long term plan of requesting follow-up events from NICOR for up to 10 years, so they can report on long term outcomes of drug coated balloon treatment.

ELIGIBILITY:
Inclusion Criteria:

All patients who were treated with drug coated balloon angioplasty during 01/01/2009 - 31/12/2015 at Norfolk and Norwich University Hospital.

-

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All comers, real life patients
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-09-11 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events (MACE) defined as a composite of all cause death, myocardial infarction and target vessel revascularisation for 12 months and then up to 10 years | 12 months and then up to 10 years
  Death. All cause death will be defined as death due to any cause.
  . Target vessel revascularisation (TVR) A TVR is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel. The latter is defined as the entire major coronary vessel proximal and distal to the target lesion, including upstream and downstream branches and the target lesion itself.
Myocardial Infarction (MI) | 12 months and then up 10 years
  An MI is defined as an episode of chest pain with positive cardiac enzyme troponin as per MINAP definition (a hospital diagnosis reported as a troponin positive MI).
Target Vessel Revascularisation (TVR) | 12 months and then up to 10 years
  A TVR is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel. The latter is defined as the entire major coronary vessel proximal and distal to the target lesion, including upstream and downstream branches and the target lesion itself.

SECONDARY OUTCOMES:
Acute vessel closure and target lesion revascularisation for 12 months and then up to 10 years. | 12 months and then up to 10 years
  Acute Vessel Closure Acute vessel closure is defined as an event where a patient had to be taken back to cardiac catheterisation lab and require repeat angioplasty (during the same hospital stay) for a complete or partial occlusion of the artery due to a dissection.
  TLR A TLR is defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion. The target lesion is defined as the treated segment from 5 mm proximal and 5 mm distal to the treated lesion (by visual assessment).
TLR | 12 months and then up to 10 years
  A TLR is defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion. The target lesion is defined as the treated segment from 5 mm proximal and 5 mm distal to the treated lesion (by visual assessment).

CONTACTS AND LOCATIONS:
Overall Officials: Upul Wickramarachchi, Dr, Principal Investigator — Norfolk & Norwich University Hospital
Locations (1):
- Norfolk and Norwich University Hospital, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Merinopoulos I, Corballis N, Gunawardena T, Bhalraam U, Natarajan R, Reinhold J, Wickramarachchi U, Maart C, Sawh C, Sulfi S, Gilbert T, Wistow T, Ryding A, Vassiliou VS, Eccleshall SC. Assessment of Scoring Balloons in STEMI Patients Treated With DCB-Only Angioplasty: A Single Center Study. Health Sci Rep. 2025 May 21;8(5):e70839. doi: 10.1002/hsr2.70839. eCollection 2025 May. PMID 40406647
- [Derived] Merinopoulos I, Gunawardena T, Corballis N, Bhalraam U, Reinhold J, Wickramarachchi U, Maart C, Gilbert T, Richardson P, Sulfi S, Sarev T, Sawh C, Wistow T, Ryding A, Mohamed MO, Perperoglou A, Mamas MA, Vassiliou VS, Eccleshall SC. Assessment of Paclitaxel Drug-Coated Balloon Only Angioplasty in STEMI. JACC Cardiovasc Interv. 2023 Apr 10;16(7):771-779. doi: 10.1016/j.jcin.2023.01.380. PMID 37045498